CLINICAL TRIAL: NCT02777931
Title: A Multicenter, 6-week, Double-blind, Randomized, Placebo-controlled, Parallel-design Study to Assess the Efficacy and Safety of NFC-1 in Adolescents (Ages 12-17) With Genetic Disorders Impacting Metabotropic Glutamate Receptors and ADHD
Brief Title: Efficacy and Safety of NFC-1 in Adolescents With Genetic Disorders Impacting mGluR and ADHD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Aevi Genomic Medicine, LLC, a Cerecor company (Industry)
Responsible Party: Sponsor
Organization: Avalo Therapeutics, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MDGN-NFC1-ADHD-201
Record Dates: First submitted 2016-05-13; First posted 2016-05-19 (Estimated); Results first posted 2018-03-29 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2018-03

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NFC-1 (Experimental): Doses of NFC-1 will be administered as 100, 200, or 400 mg twice daily as capsules for oral administration.
  Interventions: Drug: NFC-1
- Placebo (Placebo Comparator): Matching placebo capsules.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NFC-1 — NFC-1 is supplied as size 2 hard gelatin capsules.
  Other Names: NFC1
  Arms: NFC-1
Drug: Placebo — Matching placebo capsules
  Other Names: Control
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group study of NFC-1 versus placebo in adolescents with ADHD who have genetic disorders impacting mGluRs.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-group study of adolescents with ADHD who have genetic disorders impacting mGluRs. Approximately 90 subjects will receive randomized treatment with NFC-1 or placebo. Dosing will be optimized during the first 4 weeks of treatment, based on clinical response and tolerability, and maintained for an additional 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Subject has ADHD as defined by the Diagnostic and Statistical Manual of Mental Disorders, 5th edition (DSM-5) and Version 5 of the Attention Deficit Hyperactivity Disorder Rating Scale (ADHD-RS-5) ≥ 28 at Baseline with or without conventional ADHD therapy.
* Subject has an intelligence quotient (IQ) > 79, based on the Wechsler Abbreviated Scale of Intelligence, second edition (WASI-II).
* Subject has been genotyped previously and determined to have disruptive mutations in genes within the glutamate receptor metabotropic (GRM)-network as determined by the presence of copy number variations (CNVs) (GRM biomarker-positive subjects). The confirmation of a subject's positive status will be provided by the sponsor.
* Subject is judged to be in general good health, other than having ADHD, based on medical history, physical examination, vital signs measurements, laboratory safety tests, and the Columbia Suicide Severity Rating Scale (C-SSRS) performed at the Screening Visit and/or prior to administration of investigational product (IP).
* Subject has no clinically significant abnormality on electrocardiogram (ECG) performed at the Screening Visit and/or prior to administration of IP such as serious arrhythmia, bradycardia, tachycardia, cardiac conduction problems, or other abnormalities deemed to be a potential safety issue.
* Parent/legal guardian and subject understand the study procedures and agree to the subject's participation in the study as indicated by parental/legal guardian signature on the subject informed consent form and subject signature on the assent form.

Exclusion Criteria:

* Subjects with prior diagnosis of comorbid major psychiatric disorders (ie, aside from ADHD), including major depression, bipolar disease, schizophrenia, pervasive development disorder, and intellectual disability.
* Subject is currently taking a prohibited medication and/or is unwilling to wean off current ADHD medication to participate in the study
* Subject has a history of any illness that in the opinion of the study investigator might confound the results of the study or poses an additional risk to the subject by his or her participation in the study.
* Subject has a known history or presence of syncope, cardiac conduction problems (eg, clinically significant heart block), exercise-related cardiac events including syncope and pre-syncope, or clinically significant bradycardia.
* Subject has a history of stroke, chronic seizures, or major neurological disorder which, in the opinion of the investigator, would interfere with the subject's ability to participate and/or be evaluated in the study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2016-06; Primary Completion 2017-02-10 (Actual); Study Completion 2017-02-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Clinical Trials Center at Kennedy Krieger Institute, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Glessner JT, Khan ME, Chang X, Liu Y, Otieno FG, Lemma M, Slaby I, Hain H, Mentch F, Li J, Kao C, Sleiman PMA, March ME, Connolly J, Hakonarson H. Rare recurrent copy number variations in metabotropic glutamate receptor interacting genes in children with neurodevelopmental disorders. J Neurodev Disord. 2023 Apr 29;15(1):14. doi: 10.1186/s11689-023-09483-z. PMID 37120522
- [Derived] Slaby I, Hain HS, Abrams D, Mentch FD, Glessner JT, Sleiman PMA, Hakonarson H. An electronic health record (EHR) phenotype algorithm to identify patients with attention deficit hyperactivity disorders (ADHD) and psychiatric comorbidities. J Neurodev Disord. 2022 Jun 11;14(1):37. doi: 10.1186/s11689-022-09447-9. PMID 35690720

RESULTS

PARTICIPANT FLOW:
Groups:
- NFC-1: Doses of NFC-1 will be administered as 100, 200, or 400 mg twice daily as capsules (size 2 hard gelatin capsules).
Period: Overall Study
Arm/Group | NFC-1 | Placebo
Started (All randomized subjects (Intent to Treat Population)) | 49 | 52
Safety Population (All randomized subjects who took at least 1 dose of study drug) | 47 | 50
Modified Intent to Treat Population (Subjects who took at least 1 dose of study drug and have valid baseline and post baseline assessment) | 46 | 50
Completed | 37 | 39
Not Completed | 12 | 13

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | NFC-1 | Placebo | Total
Number analyzed (Participants) | 47 | 50 | 97
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.8 (1.40) | 14.4 (1.68) | 14.1 (1.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 15 | 36
  Male | 26 | 35 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 18 | 29
  White | 29 | 26 | 55
  More than one race | 6 | 3 | 9
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 47 | 50 | 97

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Attention Deficit Hyperactivity Disorder Rating Scale, Version 5 (ADHD-RS-5) Total Score
Description: The ADHD-RS-5 is comprised of 18 frequency items and 12 impairment items. Each frequency item was scored on a scale from 0 = "Never or rarely" to 3 = "Very often".
  The ADHD-RS-5 total score was calculated as the sum of the 18 frequency item scores. The total score ranges from 0 to 54. Higher scores indicate greater symptom severity. Change from baseline value were calculated as the assessment value minus the baseline value.
Time Frame: Baseline to Visit 8 (Week 6)
Population: Modified Intent to Treat Population = all randomized subjects who took at least one dose of randomized study drug and have a valid baseline assessment and at least 1 valid post baseline assessment.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NFC-1 | Placebo
Number analyzed (Participants) | 46 | 50
units on a scale | -14.2 (1.82) | -12.1 (1.75)

2. Primary Outcome: Clinical Global Impression - Global Improvement (CGI -I) Response
Description: The CGI-I item is rated on a 7-point scale from 1 = "Very much improved", 2 = "Much improved", 3 = "Minimally improved", 4 = "No change", 5 = "Minimally worse", 6 = "Much worse", 7 = "Very much worse".
  Response is defined as achieving a CGI-I score of 1 or 2, scores of 3 to 7 or missing are defined as Non Response
Time Frame: Visit 3 to Visit 8 (Week 6)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | NFC-1 | Placebo
Number analyzed (Participants) | 46 | 50
Participants | 26 | 16

ADVERSE EVENTS:
Time Frame: 8 months, 5 days
Arm/Group | NFC-1 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/50
Other Adverse Events (participants affected / at risk) | 33/47 | 28/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NFC-1 (N=47) | Placebo (N=50)
Nausea (Gastrointestinal disorders) | 3 (3) | 4 (4)
Fatigue (General disorders) | 7 (7) | 3 (3)
Nasopharyngitis (Infections and infestations) | 1 (1) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 5 (5)
Accidental overdose (Injury, poisoning and procedural complications) | 5 (7) | 3 (3)
Weight increase (Investigations) | 7 (7) | 2 (2)
Increased appetite (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 4 (5) | 5 (10)
Irritability (Psychiatric disorders) | 1 (1) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The information generated by this study is the property of Medgenics. Publication or other public presentation of NFC-1 data resulting from this study requires prior review and written approval of Medgenics. Abstracts, manuscripts, and presentation materials should be provided to Medgenics for review at least 30 days prior to the relevant submission deadline.

DOCUMENTS (2):
  • Study Protocol (2016-10-27): https://cdn.clinicaltrials.gov/large-docs/31/NCT02777931/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-30): https://cdn.clinicaltrials.gov/large-docs/31/NCT02777931/SAP_001.pdf